CLINICAL TRIAL: NCT02000102
Title: Outcomes of Diabetic Macula Edema Patients Switched to Aflibercept From Bevacizumab and/or Ranibizumab
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 28279
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Diabetic Macular Edema Patients Switched to Aflibercept
  Interventions: Drug: Intravitreal Injection of Aflibercept

INTERVENTIONS:
Drug: Intravitreal Injection of Aflibercept

SUMMARY:
Patients with diabetic macular edema who were switched to aflibercept after having been treated with bevacizumab or ranibizumab were retrospectively reviewed to assess for visual acuity and anatomic outcomes.

ELIGIBILITY:
Inclusion Criteria: Those patients with diabetic macular edema switched to aflibercept from bevacizumab and/or ranibizumab -

Exclusion Criteria: None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients with diabetic macular edema switched to aflibercept from bevacizumab and/or ranibizumab
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 1 year

SECONDARY OUTCOMES:
Central Subfield Thickness on Optical Coherence Tomography | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States